CLINICAL TRIAL: NCT07190521
Title: Hypnobreastfeeding vs. Traditional Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Merve İrem İslikaye
Record Dates: First submitted 2025-07-18; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Prenatal Education Group Hypnobreastfeeding Group
  Interventions: Other: hypnobreastfeeding education; Other: Traditional prenatal education
- Control group (No Intervention): Control Group

INTERVENTIONS:
Other: hypnobreastfeeding education — Hypnobreastfeeding education is an antenatal training method that combines:
  Hypnotherapy principles
  Guided imagery
  Affirmations
  Breathing and deep relaxation techniques
  Arms: intervention group
Other: Traditional prenatal education — Traditional prenatal education programs, often referred to as antenatal or maternity school classes, are structured group sessions provided to pregnant women, typically in clinical or community settings. These classes aim to:
  Prepare expectant mothers for labor, birth, and postpartum care,
  Provide evidence-based information about breastfeeding, newborn care, and maternal recovery,
  Promote positive health behaviors during pregnancy,
  Reduce fear and anxiety by increasing knowledge and confidence.
  Arms: intervention group

SUMMARY:
Breastfeeding is a vital component of maternal and infant health, and its success is closely linked to the mother's psychological readiness, self-efficacy, and perception of milk sufficiency. In recent years, alternative educational approaches such as hypnobreastfeeding, which integrates hypnosis and relaxation techniques into prenatal education, have gained increasing attention. These approaches aim to improve maternal self-efficacy, reduce stress and anxiety during the breastfeeding period, and promote better adaptation to breastfeeding in the early postpartum phase.

Traditional prenatal breastfeeding education primarily focuses on anatomical, physiological, and practical aspects of breastfeeding. While effective, this approach may not sufficiently address maternal fears, emotional barriers, or negative birth experiences that can undermine breastfeeding outcomes.

In contrast, hypnobreastfeeding education incorporates guided imagery, affirmations, breathing techniques, and deep relaxation, offering a more holistic preparation for breastfeeding. Emerging studies suggest that mothers who receive hypnobreastfeeding training demonstrate higher levels of breastfeeding self-efficacy, stronger emotional bonding, better adaptation to breastfeeding, and lower perceptions of insufficient milk compared to those receiving standard education.

This review explores the comparative effectiveness of hypnobreastfeeding versus traditional prenatal breastfeeding education, focusing on three key outcomes: maternal self-efficacy, breastfeeding adaptation, and perceived insufficient milk supply. The findings indicate that combining psychological readiness techniques with conventional education may enhance maternal confidence and breastfeeding continuity.

Further research with larger sample sizes and long-term follow-up is needed to validate the integration of hypnobreastfeeding into routine antenatal care.

DETAILED DESCRIPTION:
Prenatal Education Group:

Traditional prenatal education programs provide information-based training on childbirth and newborn care, including breastfeeding. This method is primarily knowledge-focused and offers mothers guidance on breastfeeding techniques, common problems, and suggested solutions.

Hypnobreastfeeding Group:

This method aims to help mothers develop relaxation, self-confidence, and stress management skills regarding breastfeeding through the use of hypnosis techniques. Hypnosis may support mothers in forming more positive subconscious beliefs about breastfeeding.

Control Group:

All first-time pregnant mothers who do not receive either traditional prenatal education or hypnobreastfeeding training will be included in this group.

ELIGIBILITY:
Inclusion Criteria:

Gestational age between 28 and 36 weeks,

Primiparous pregnant women,

Age between 18 and 40 years,

Singleton pregnancy,

Spontaneous conception (not assisted reproductive technology),

No visual or hearing impairments,

No communication difficulties,

Completion of traditional prenatal (antenatal) education,

Completion of hypnobreastfeeding education,

No medical conditions preventing breastfeeding (e.g., anatomical breast issues),

Voluntary participation in the study.

Exclusion Criteria Diagnosis of high-risk pregnancy,

Multiple pregnancy (twins, triplets, etc.),

Conception via assisted reproductive techniques,

Diagnosis of a severe psychiatric disorder,

Failure to complete either prenatal education or hypnobreastfeeding education,

Declining to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnacy
Enrollment: 111 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
To determine the breastfeeding self-efficacy levels of mothers. | 16 weeks
  Assessed using the Breastfeeding Self-Efficacy Scale
To determine the breastfeeding Adaptation levels of mothers. | 16 weeks
  (Assessed using the Breastfeeding Adaptation Scale.)

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For ethical reasons, patient information may be shared upon reasonable request without revealing their identities for security reasons.